CLINICAL TRIAL: NCT00805922
Title: DiabCare Asia 2008. A Cross-Sectional Survey to Evaluate Diabetes Management, Control, Complications, Psychosocial Aspects of Diabetic Patients in Asia and To Evaluate Perceptions and Practices of Physicians and Patients About Diabetes Management in Asia
Brief Title: A Survey to Evaluate Diabetes Management, Control, Chronic Complications, Psychosocial Aspects of Diabetic Subjects in Thailand
Acronym: DiabCare Asia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3707
Record Dates: First submitted 2008-12-09; First posted 2008-12-10 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Capillary or venous blood will be drawn for analysing HbA1c.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Capillary or venous blood will be drawn for analysing HbA1c.

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate current status of diabetes management, control, complications in diabetic subjects in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients registered in the particular centre for more than 12 months.
* Patients should have visited the centre at least once in the last 3-6 months apart from the initial visit.
* Patients willing to sign informed consent form.

Exclusion Criteria:

* Repetition of any patient as patients should not be included twice for any reason.
* Unwilling to participate or unable to comply with protocol requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus being treated at general hospitals, diabetes clinics and referral clinics will be selected according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2342 (Actual)
Dates: Start 2008-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean blood glucose parameters of diabetic patients | Study start

SECONDARY OUTCOMES:
Patients' perception will be analysed through patient questionnaire measuring psychological well-being, quality of life and patients' compliant to treatment | Study start
Physician perception of diabetes and its management will be analysed through physician questionnaire measuring awareness about HbA1c test and its goal, anti-diabetic treatment and barriers towards optimum diabetes control | Study start
Duration of diabetes associated with highest number of diabetic complications | Study start
Minimum duration of diabetes associated with 10% incidence of diabetic complications (CVD, Nephropathy and retinopathy) | Study start

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangkok, Thailand

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com